CLINICAL TRIAL: NCT02084355
Title: Efficacy and Safety of Opioid Rotation Compared With Opioid Dose Escalation in Patients With Moderate to Severe Cancer Pain - Open Label, Randomized, Prospective Study
Brief Title: Study of Opioid Rotation Versus Opioid Escalation in Patients With Moderate to Severe Cancer Pain
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Gyeongsang National University Hospital (Other)
Responsible Party: Principal Investigator, Jung Hun Kang, Associate Professor, Gyeongsang National University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: GNUH-2013-07-014
Record Dates: First submitted 2014-03-05; First posted 2014-03-12 (Estimated); Last update posted 2014-03-12 (Estimated); Status verified 2014-03

CONDITIONS: Cancer; Pain
Keywords: Significant cancer pain; at least numeric rating scale 4
MeSH Terms: conditions — Neoplasms; Pain | interventions — Oxycodone; Hydromorphone

ARMS (2):
- opioid rotation (Experimental): Patients who are randomized to opioid rotation are treated with strong opioid other than currently used strong opioid (Reduce the dose by 25%-50% to allow for incomplete cross-tolerance between different opioids).
  * oral oxycodone : convert to oral hydromorphone or fentanyl patch
  * oral hydromorphone : convert to oral oxycodone or fentanyl patch
  * fentanyl patch : convert to oral oxycodone or oral hydromorphone
  Interventions: Drug: oral oxycodone; Drug: oral hydromorphone; Drug: fentanyl patch
- opioid dose escalation (Active Comparator): Patients who are randomized to opioid dose escalation will be treated cancer pain by escalation dose of same strong opioid.
  * oral oxycodone : maintain oral oxycodone and titrate the dose
  * oral hydromorphone : maintain oral hydromorphone and titrate the dose
  * fentanyl patch : maintain fentanyl patch and titrate the dose
  Interventions: Drug: oral oxycodone; Drug: oral hydromorphone; Drug: fentanyl patch

INTERVENTIONS:
Drug: oral oxycodone
Drug: oral hydromorphone
Drug: fentanyl patch

SUMMARY:
Although opioid rotation is well known treatment modality in reducing pain and opioid-induced neurotoxicity, it is not established whether opioid rotation is more appropriate or opioid escalation is more effective in controlling significant pain in cancer patients under opioid medication.

- The purpose of this study is to determine effective therapy out of opioid rotation and opioid dose escalation in patients with moderate to severe cancer pain who have been already treated with strong opioid.

ELIGIBILITY:
Inclusion Criteria:

* age > 18 years
* patients who are being treated with one of strong opioids including oral oxycodone, oral hydromorphone, or fentanyl patch with range from 60 mg to 200 mg of oral morphine equivalent daily dose (MEDD)
* moderate to severe cancer pain (numeric rating scale more than 3) at screening
* patients without uncontrolled adverse effects associated with currently applied opioid

Exclusion Criteria:

* previous opioid rotation
* unable to take oral medication
* life expectancy less than a month
* newly started chemotherapy and/or radiotherapy within past 2 weeks of screening
* serum aspartate aminotransferase, alanine aminotransferase, or alkaline phosphatase > 2.5 times of upper normal limit
* serum total bilirubin or creatinine > 1.5 times of upper normal limit

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 136 (Estimated)
Dates: Start 2014-04; Primary Completion 2015-12 (Estimated); Study Completion 2016-01 (Estimated)

PRIMARY OUTCOMES:
The rate of successful pain control defined as a 30% or 2-point reduction in the numeric rating scale | Eighteen months

CONTACTS AND LOCATIONS:
Locations (1):
- Gyeongsang National University Hospital, Jinju, Gyeongsangnam-do, South Korea